CLINICAL TRIAL: NCT06959498
Title: Long-term Survival of THA After Pelvic and/or Femoral Osteotomy
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Olivier ROCHE, Dr, Central Hospital, Nancy, France
Other Study IDs: 2024PI083
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Hip Arthropathy Associated With Other Conditions; Hip Dysplasia; Survival, Prosthesis
MeSH Terms: conditions — Hip Dislocation; Prosthesis Failure | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pelvic osteotomy or shelf acetabuloplasty: Total hip arthroplasty after pelvic osteotomy or shelf acetabuloplasty
  Interventions: Procedure: Total hip arthroplasty
- Femoral osteotomy: Total hip arthroplasty after femoral osteotomy
  Interventions: Procedure: Total hip arthroplasty
- Combined osteotomy: Total hip arthroplasty after a combination of pelvic osteotomy or shelf acetabuloplasty, and femoral osteotomy
  Interventions: Procedure: Total hip arthroplasty

INTERVENTIONS:
Procedure: Total hip arthroplasty — Total hip arthroplasty

SUMMARY:
Analyze the long-term clinical and radiological outcomes of total hip arthroplasty (THA) in patients with hip dysplasia treated by pelvic osteotomy, femoral osteotomy, shelf acetabuloplasty, or a combination of these interventions, performed during childhood or early adulthood. The aim is to understand the impact of these early interventions on THA survival and long-term joint function.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent THA between 1998 and 2010 and had a prior surgical treatment for hip dysplasia (pelvic, femoral osteotomy, shelf acetabuloplasty or combined osteotomy)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients, with no age limit, operated in the Centre Chirurgical Emile Gallé, Nancy, France, between 1998 and 2010
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
survival | 20 years
  Study of 15 year survival of THA